CLINICAL TRIAL: NCT00939939
Title: Effect of Sitagliptin on Postprandial Lipoprotein Metabolism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Prof. Klaus Parhofer, Med. Dept. 2 University Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP MSD 01-08
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitagliptin (Experimental)
  Interventions: Drug: sitagliptin
- glimepirid (Active Comparator)
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: sitagliptin — sitagliptin 100 mg/d for 10 weeks
  Arms: sitagliptin
Drug: glimepiride — glimepiride 1 mg/d for 10 weeks
  Arms: glimepirid

SUMMARY:
The goal of the study is to evaluate whether sitagliptin can affect postprandial lipoprotein metabolism in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* dietary therapy

Exclusion Criteria:

* lipid-lowering therapy
* anti-hyperglycemic drug therapy

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
incremental area under the triglyceride curve (iAUC-TG) | 10 weeks
  incremental area under the plasma triglyceride concentration curve following a standardized oral fat challenge

SECONDARY OUTCOMES:
LDL-cholesterol | 10 weeks
  fasting LDL-cholesterol
HDL-cholesterol | 10 weeks
  fasting HDL-cholesterol
VLDL-cholesterol | 10 weeks
  fasting VLDL-cholesterol
triglycerides | 10 weeks
  fasting triglycerides
area under the triglyceride curve (AUC-TG) | 10 weeks
  area under the plasma triglyceride concentration curve following a standardized oral fat challenge
area under the VLDL-triglyceride curve (AUC-VLDL-TG) | 10 weeks
  area under the plasma VLDL-triglyceride concentration curve following a standardized oral fat challenge
incremental area under the VLDL-triglyceride curve (iAUC-VLDL-TG) | 10 weeks
  incremental area under the plasma VLDL-triglyceride concentration curve following a standardized oral fat challenge
glucose | 10 weeks
  fasting glucose concentration
insulin | 10 weeks
  fasting insulin concentration
HOMA | 10 weeks
HbA1c | 10 weeks
interleukin-6 | 10 weeks
hs-CRP | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Dept. 2, Grosshadern, University Munich, Munich, Germany